CLINICAL TRIAL: NCT02226718
Title: Validation of a Questionnaire for Measuring Health-related Quality of Life in Patients With Chronic Otitis Media
Brief Title: Validation of a Questionnaire for Measuring Quality of Life in Patients With Chronic Inflammation of the Middle Ear
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: HRQOL-COM1
Record Dates: First submitted 2014-08-14; First posted 2014-08-27 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Chronic Otitis Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- questionnaire: Otitis patients and controls
  Interventions: Other: Administration of questionnaire

INTERVENTIONS:
Other: Administration of questionnaire

SUMMARY:
For measuring quality of life in patients with chronic inflammation of the middle ear, only two questionnaires currently exist. However, these questionnaires are designed only to measure either disease-specific health or hearing-related quality of life. The aim of this project is the validation of a pre-existing comprehensive questionnaire, which is routinely administered in the investigators clinic but has never been validated. Following a retrospective item reduction based on existing data, this questionnaire will be prospectively validated. Applying the resulting questionnaire in future studies on chronic middle ear inflammation, not only objective outcome parameters (e.g. audiograms) but also quality of life will be assessed. Therefore, the investigators questionnaire will add substantial information to these outcome studies by providing a subjective outcome parameter.

DETAILED DESCRIPTION:
See Summary that contains all the details

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of chronic otitis media

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffering from chronic otitis media, visiting a tertiary referral centre
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Validity | day 1 (day of consultation)
  Several aspects of Validity will be determined by different methods:
  * content validity is made certain by construction procedure of the questionnaire (e.g. involving of specialists and patients)
  * construct validity by factor analysis
  * criterion validity by correlating a global question with the overall questionnaire score

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Huber, M.D., Principal Investigator — Universitätsspital Zürich
Locations (1):
- Universitätsspital Zürich, Zurich, Switzerland